CLINICAL TRIAL: NCT00406562
Title: Open, Booster Vaccination Study to Assess Safety and Reactogenicity of GSK Biologicals' dTpa Vaccine (Boostrix) When Administered to Healthy Chinese Children 6-8 Years of Age.
Brief Title: Study to Assess the Safety & Reactogenicity of GSK Biologicals' dTpa Vaccine (Boostrix) When Given at 6-8 Years of Age.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 107924
Record Dates: First submitted 2006-12-01; First posted 2006-12-04 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Tetanus; Diphtheria; Acellular Pertussis
Keywords: uncontrolled
MeSH Terms: conditions — Tetanus; Diphtheria | interventions — Boostrix

INTERVENTIONS:
Biological: Boostrix

SUMMARY:
This study will evaluate the safety and reactogenicity of booster dose of GSK Biologicals' dTpa vaccine (Boostrix) in Chinese children at 6-8 years of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between, and including, 6-8 years of age at the time of vaccination,
* Written informed consent obtained from the parent or guardian of the subject,
* Subjects who have received a total of 4 doses of DTP vaccine in the first 2 years of life,

Exclusion Criteria:

* subjects who have received previous DTP booster vaccination since administration of the fourth dose of vaccine in second year of life can not participate
* Subjects with history of diphtheria, pertussis or tetanus diseases can not participate

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30
Dates: Start 2007-01; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited symptoms during 4 days following vaccination, unsolicited symptoms during the 31 days following vaccination and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Suining, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Zhu F, Zhang S, Hou Q, Zhang Y, Xu Y, Ma X, Lu X, Pan H, Chen D, Ramakrishnan G, Zhao R, Tang H, Van Der Meeren O, Bock HL. Booster vaccination against pertussis in Chinese children at six years of age using reduced antigen content diphtheria-tetanus-acellular pertussis vaccine (Boostrix()). Hum Vaccin. 2010 Mar 3;6(3):10503. doi: 10.4161/hv.6.3.10503. Epub 2010 Mar 3. PMID 20215881
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 107924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register